CLINICAL TRIAL: NCT02619435
Title: Regorafenib Monotherapy as Second-line Treatment of Patients With RAS-mutant Advanced Colorectal Cancer: a Multicentre, Single-arm, Two-stage, Phase 2 Study
Brief Title: Regorafenib Monotherapy as Second-line Treatment of Patients With RAS-mutant Advanced Colorectal Cancer
Acronym: STREAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STREAM; 2015-001105-13 (EudraCT Number)
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Advanced Colorectal Cancer
Keywords: RAS-mutant
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- regorafenib (Experimental)
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — Patients will receive regorafenib orally 160 mg once daily for the first 3 weeks of each 4-week cycle.

SUMMARY:
The purpose of this study is to purpose of this study is to assess if regorafenib is active enough, in terms of 6-month progression-free rate, to warrant further comparative studies in patients with RAS-mutant advanced colorectal cancer who have progressed after first-line oxaliplatin-based chemotherapy plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of colorectal adenocarcinoma
2. Any RAS mutation that prevent treatment with anti-EGFR antibodies
3. Stage IV
4. Measurable disease according to RECIST v. 1.1
5. Disease progression during or following a treatment with fluoropyrimidine, oxaliplatin and bevacizumab, and a treatment with irinotecan is not considered immediately mandatory by the Investigator
6. Age ≥ 18 years
7. ECOG Performance Status 0-1
8. Neutrophils > 1500 / mm3, platelets > 100,000 / mm3, and hemoglobin > 9 g/dL without transfusion or granulocyte-colony stimulating factor (G-CSF) and other hematopoietic growth factors.
9. Bilirubin level < 1.5 x ULN
10. Glomerular filtration rate > 30 mL/min/1.73 m2 according to the Modified Diet in Renal Disease abbreviated formula
11. AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN (≤ 5 x ULN if liver metastasis are present)
12. Alkaline phosphatase ≤ 2.5 x ULN (≤ 5 x ULN if liver metastasis are present)
13. Serum creatinine < 1.5 x ULN
14. Amylase and lipase ≤ 1.5 x ULN
15. INR and aPTT ≤ 1.5 x ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no underlying abnormality in coagulation parameters exists per medical history.
16. Understand, be willing to give consent, and sign the written informed consent form (ICF) prior to undergoing any study-specific procedure.
17. If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment.
18. If potentially childbearing female, or if male, agree to use adequate contraception (eg, abstinence, intrauterine device, oral contraceptive, or double-barrier method) from the date on which the ICF is signed until 8 weeks after the last dose of study drug.
19. Life expectancy of greater than 3 months

Exclusion Criteria:

1. Previous treatment with regorafenib or irinotecan
2. Are taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort)
3. Have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment
4. Have congestive heart failure classified as New York Heart Association Class 2 or higher
5. Have had unstable angina (angina symptoms at rest) or new-onset angina < 3 months prior to screening.
6. Have had a myocardial infarction < 6 months prior to initiation of study treatment.
7. Have cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin.
8. Have had arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months prior to the initiation of study treatment
9. Symptomatic brain metastases or meningeal tumors
10. Patients with evidence or history of bleeding diathesis
11. Uncontrolled hypertension (systolic blood pressure [SBP] >140 mmHg or diastolic blood pressure [DBP] > 90 mmHg)
12. Have interstitial lung disease with ongoing signs and symptoms at the time informed consent is obtained
13. Have persistent proteinuria > 3.5 g/24 hours measured by urine protein creatinine ratio from a random urine sample (< Grade 3, CTCAE v 4.0).
14. Have unresolved toxicity higher than National Cancer Institute-Common Terminology for Adverse Events version 4.0 (CTCAE v 4.0) Grade 1 attributed to any prior therapy/procedure, excluding alopecia and/or oxaliplatin-induced neurotoxicity ≤ Grade 2 and hemoglobin ≥ 9 g/dL as per inclusion criteria
15. Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease
16. Pregnant or lactating women
17. Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or non melanoma skin cancer)
18. Any unstable systemic disease (including active infections, any significant hepatic, renal or metabolic disease), metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of regorafenib or render the patient at high risk for treatment complications
19. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
20. Have any other serious or unstable illness, or medical, psychological, or social condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results.
21. Have a known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs.
22. Have a close affiliation with the investigational site (eg, be a close relative of the investigator) or be a dependent person (eg, be an employee or student working at the investigational site).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2015-11; Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
the rate of evaluable patients alive and not progressed at 6 months | 6 months

SECONDARY OUTCOMES:
worst grade toxicity per patient | every 4 weeks up to 1 year
  evaluated according to RECIST 1.1
number of patients with complete plus partial response | 6 months
progression free survival | up to one year
  the time from registration to progression or death without progression
overall survival | up to 2 years
  as the time from registration to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Avallone, M.D., Principal Investigator — National Cancer Institute, Naples; Alfredo Budillon, M.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (4):
- Italy (4):
  - AO G. Rummo, Benevento
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Seconda Università di Napoli, Napoli
  - AO S. Carlo, Potenza